CLINICAL TRIAL: NCT06620757
Title: Safety and Effectiveness of Short-Term Single AntiPlatelet Therapy After Left Atrial Appendage Closure With the LAmbre Device in Patients With Nonvalvular Atrial Fibrillation: A Multinational Real-world Registry
Acronym: S-SAPT LAMBRE
Status: Recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC39-S-SAPT LAMBRE
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage Closure; Single Antiplatelet Therapy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Antiplatelet therapy after Left Atrial Appendage Occlusion (LAAO)
  Interventions: Drug: Single antiplatelet therapy (SAPT)

INTERVENTIONS:
Drug: Single antiplatelet therapy (SAPT) — Observational study of effectiveness and safety of SAPT (either with acetyl-salycilic acid or clopidogrel) after LAAO with Lambre device in patients with high risk of bleeding

SUMMARY:
Brief Summary: A prospective, multicenter, single-arm, non-randomized study including consecutive patients with nonvalvular AF(Atrial Fibrillation), with a CHA2DS2-VASc score ≥2 (men) or ≥3 (women), and contraindication for long-term anticoagulant treatment, with successful LAAC (Left Atrial Appendage Closure)procedure with the LAmbre device, who at discharge are eligible for short-term (3-months-only) SAPT. We want to assess if a short-term single antiplatelet therapeutic regime of Acetylsalicylic acid (ASA) 100 mg (or clopidogrel 75 mg if ASA contraindication), once daily, for 3 months is safe and effective at 12 months follow-up.

DETAILED DESCRIPTION:
The S-SAPT SECURE-LAMBRE REGISTRY is a prospective, multicenter, single-arm, non-randomized study including consecutive patients with nonvalvular AF, with a CHA2DS2-VASc score ≥2 (men) or ≥3 (women), and contraindication for long-term anticoagulant treatment, with successful LAAC procedure with the LAmbre device, who at discharge are eligible for short-term (3-months-only) SAPT.

234 patients will be enrolled in the study. The study will be conducted at about 20 investigational centers in Spain. The enrollment phase is expected to take approximately 18 months.

Patients included in the study will be clinically followed for 12 months. In addition patients will have imaging (TEE or cCT) follow-up at 45-90 days and 12 month.

The hypothesis of the study is the following: After successful procedure of implantation of the Lifetech LAmbre Left Atrial Appendage Closure (LAAC) device in patients with nonvalvular paroxysmal, persistent, or permanent Atrial Fibrillation (AF), a short-term single antiplatelet therapeutic regime of Acetylsalicylic acid (ASA) 100 mg (or clopidogrel 75 mg if ASA contraindication), once daily, for 3 months is safe and effective at 12 months follow-up.

Objectives:

Primary objective. To evaluate the occurrence of stroke and thromboembolic events at 12 months with short-term SAPT with ASA 100 mg (or clopidogrel 75 mg if ASA contraindication) once daily during 3 months after successful LAAC with the LAmbre device.

Secondary objective. To evaluate the occurrence of major bleeding events at 12 months with short-term SAPT with ASA 100 mg (or clopidogrel 75 mg if ASA contraindication) during 3 months after successful LAAC with the LAmbre device.

Endpoints:

Primary endpoint. A composite of stroke (including ischemic and/or hemorrhagic) and/or systemic embolism at 12 months.

Secondary endpoints.

1. Device thrombosis at 45-90 days, if suggested by Transesophageal Echocardiography (TEE), confirmed by a cardiac Computed Tomography (cCT) scan.
2. Device thrombosis at 1 year, if suggested by TEE, confirmed by a CT scan.
3. Cardiovascular death at 12 months.
4. Nonprocedural major bleeding events (Bleeding Research Academy Consortium [BARC] ≥3b) at 12 months.
5. The composite of cardiovascular death, stroke, systemic embolism, and nonprocedural bleeding at 12 months.
6. All-cause death at 12 months. This study has an steering Committee, an independent Data and Safety Monitoring Board (DSMB) and independent Clinical Events Committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

All criteria must be met

* Patient 18 years and over and
* Patient with documented nonvalvular AF, defined as AF in the absence of moderate or severe mitral stenosis or a mechanical heart valve and
* Patient with a calculated CHA₂DS₂-VASc score ≥2 (for men) and ≥3 (for women) and
* Patient with a contraindication for long-term anticoagulant treatment and
* Patient who has undergone a successful LAmbre LAAC device implantation with no complications during the in-hospital period after the intervention and
* Patient able and willing to return for required follow-up visits and examinations and
* Patient with Informed consent signed.

Exclusion Criteria:

No exclusion criteria must be met.

* Patient is currently enrolled in another investigational study, except when the subject is participating in a purely observational registry with no associated treatments.
* Patient requires long-term anticoagulation therapy for reasons other than AFrelated stroke risk reduction, for example, due to an underlying hypercoagulable state (i.e even if the device is implanted, the subjects would not be eligible to discontinue OAC (Oral Anticoagulation) due to other medical conditions requiring chronic OAC therapy).
* Patient has contraindications or is allergic to both aspirin and clopidogrel.
* Patient has an indication for chronic aspirin or clopidogrel treatment (i.e., chronic ischemic disease or peripheral artery disease); thus, the subject would not be eligible to discontinue aspirin or clopidogrel due to other medical conditions requiring this therapy.
* Patient had or is planning to have any cardiac or noncardiac intervention or surgical procedure within 30 days before or 60 days after implant (including, but not limited to: cardioversion, PCI (Percutaneous Coronary Intervention), cardiac ablation, cataract surgery, etc.).
* Patient had a prior stroke (of any cause, whether ischemic or hemorrhagic) or transient ischemic attack (TIA) within the 30 days prior to enrollment.
* Patient had a major bleeding event within the 30 days prior to inclusion. Lack of resolution of related clinical sequelae or planned and pending interventions to resolve bleeding/bleeding source are further exclusions, regardless of the timing of the bleeding event.
* Patient has an active bleeding.
* Patient has had an MI documented in the clinical record as either a NSTEMI or STEMI, with or without intervention, within 30 days prior to enrollment.
* Patient has a history of atrial septal repair or has an ASD/PFO device.
* Patient is of childbearing potential, or plans to become pregnant during the study (method of assessment upon study physician's discretion).
* Patient had subject has a documented life expectancy of less than one year.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with nonvalvular AF, with a CHA₂DS₂-VASc score ≥2 (men) or ≥3 (women), contraindication for long-term anticoagulant treatment, with implantation procedural success of LAAC with the LAmbre device, who at discharge are eligible for short-term (3-months-only) SAPT
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite of stroke | 12 month
  A composite of stroke (including ischemic and/or hemorrhagic) and/or systemic embolism

SECONDARY OUTCOMES:
Device thrombosis | 45 days to 90 days
  Freedom from device thrombosis by Echocardiography (TEE), confirmed by a cardiac Computed Tomography (CT) scan
Device thrombosis | 12 months
  Freedom from device thrombosis by Transesophageal Echocardiography (TEE), confirmed by a cardiac Computed Tomography (CT) scan
Cardiovascular death | 12 months
  Freedom of Cardiovascular death
Major bleeding | 12 months
  Freedom from major bleeding events according to Academy Consortium [BARC] ≥3b)
Composite of cardiovascular death | 12 months
  Freedom from stroke, systemic embolism, and nonprocedural bleeding
All cause of death | 12 month
  Freedom from All cause of death

CONTACTS AND LOCATIONS:
Locations (22):
- Spain (22):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Clínico San Carlos, Aravaca
  - Hospital Del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía de Córdoba, Córdoba
  - Hospital Universitario La Paz, Fuencarral-El Pardo
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de Leon, León
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Central de La Defensa Gómez Ulla, Madrid
  - Hospital Universitario Puerta De Hierro, Majadahonda
  - Hospital de Manises, Manises
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario de Tarragona Juan XXIII, Tarragona
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Background] Krijthe BP, Kunst A, Benjamin EJ, Lip GY, Franco OH, Hofman A, Witteman JC, Stricker BH, Heeringa J. Projections on the number of individuals with atrial fibrillation in the European Union, from 2000 to 2060. Eur Heart J. 2013 Sep;34(35):2746-51. doi: 10.1093/eurheartj/eht280. Epub 2013 Jul 30. PMID 23900699
- [Background] Michaud GF, Stevenson WG. Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):353-361. doi: 10.1056/NEJMcp2023658. No abstract available. PMID 33503344
- [Background] Alkhouli M, Ellis CR, Daniels M, Coylewright M, Nielsen-Kudsk JE, Holmes DR. Left Atrial Appendage Occlusion: Current Advances and Remaining Challenges. JACC Adv. 2022 Nov 16;1(5):100136. doi: 10.1016/j.jacadv.2022.100136. eCollection 2022 Dec. PMID 38939465
- [Background] Glikson M, Wolff R, Hindricks G, et al. EHRA/EAPCI expert consensus statement on catheter-based left atrial appendage occlusion - an update. Europace 2022; 24(1): 71-164.
- [Background] Freeman JV, Higgins AY, Wang Y, Du C, Friedman DJ, Daimee UA, Minges KE, Pereira L, Goldsweig AM, Price MJ, Reddy VY, Gibson D, Doshi SK, Varosy PD, Masoudi FA, Curtis JP. Antithrombotic Therapy After Left Atrial Appendage Occlusion in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2022 May 10;79(18):1785-1798. doi: 10.1016/j.jacc.2022.02.047. PMID 35512858
- [Background] Carvalho PEP, Gewehr DM, Miyawaki IA, Nogueira A, Felix N, Garot P, Darmon A, Mazzone P, Preda A, Nascimento BR, Kubrusly LF, Cardoso R. Network Meta-Analysis of Initial Antithrombotic Regimens After Left Atrial Appendage Occlusion. J Am Coll Cardiol. 2023 Oct 31;82(18):1765-1773. doi: 10.1016/j.jacc.2023.08.010. Epub 2023 Aug 21. PMID 37611779
- [Background] Korsholm K, Nielsen KM, Jensen JM, Jensen HK, Andersen G, Nielsen-Kudsk JE. Transcatheter left atrial appendage occlusion in patients with atrial fibrillation and a high bleeding risk using aspirin alone for post-implant antithrombotic therapy. EuroIntervention. 2017 Apr 20;12(17):2075-2082. doi: 10.4244/EIJ-D-16-00726. PMID 27973336
- [Background] Park JW, Sievert H, Kleinecke C, Vaskelyte L, Schnupp S, Sievert K, Lam YY, Stahli BE, Zhang D, Li A, Brachmann J. Left atrial appendage occlusion with lambre in atrial fibrillation: Initial European experience. Int J Cardiol. 2018 Aug 15;265:97-102. doi: 10.1016/j.ijcard.2018.02.120. PMID 29885707
- [Background] Llagostera-Martin M, Cainzos M, Salvatella N, Cubero-Gallego H, Mas-Stachurska A, Sanchez-Carpintero A, Tizon-Marcos H, Calvo-Fernandez A, Molina L, Vaquerizo B. Single antiplatelet therapy after left atrial appendage closure in patients with AF: safety and effectiveness. Rev Esp Cardiol (Engl Ed). 2024 Feb;77(2):150-157. doi: 10.1016/j.rec.2023.06.020. Epub 2023 Oct 23. English, Spanish. PMID 37879431